CLINICAL TRIAL: NCT02133443
Title: Neurally Adjusted Ventilatory Assist (NAVA) Levels Titration During Weaning Using Ventilatory Comfort Scales: a Physiological Evaluation
Brief Title: NAVASET: Nava Level Titration Using Comfort Scales
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Nicolas TERZI, MD-PhD, University Hospital, Caen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-A01835-40; 2013-A01835-40 (Other: CPP Nord-Ouest III)
Record Dates: First submitted 2014-04-30; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Acute Respiratory Failure
Keywords: Mechanical ventilation; Acute respiratory failure; Weaning; Pressure support ventilation; Neurally adjusted ventilatory assist
MeSH Terms: interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pressure Support Ventilation (Active Comparator): Device: PSV - pressure support ventilation
  Interventions: Device: PSV - pressure support ventilation
- Neurally Adjusted Ventilatory Assist (Active Comparator): Device: Partial ventilator support with partial ventilation mode (NAVA)
  Interventions: Device: Neurally Adjusted Ventilatory Assist

INTERVENTIONS:
Device: PSV - pressure support ventilation — Gold standard partial ventilator support: Pressure Support Ventilation performed with Servo-i® ventilator (MAQUET,Critical Care, Sweden). Pressure support ventilator assistance to obtain a tidal volume of 6-8 ml/kg of ideal body weight.
  Arms: Pressure Support Ventilation
Device: Neurally Adjusted Ventilatory Assist — Partial ventilator support partial ventilation mode (NAVA) performed with Servo-i® ventilator (Maquet,Critical Care, Sweden). Different levels of neurally adjusted ventilatory assist are tested. Stepwise implementation of the NAVA level (steps of 25% ), returning to the " optimal " level between each evaluation (PSV 100%, NAVA 100%, 75%, 50%, 125%, 150%).
  Arms: Neurally Adjusted Ventilatory Assist

SUMMARY:
Determining the optimal Neurally Adjusted Ventilatory Assist (NAVA) level remains challenging, and several methods have been suggested. However none of them seems easily utilisable. Thus the investigators propose to test a way of NAVA level titration according to ventilator comfort.

DETAILED DESCRIPTION:
Physiological comparison of different levels of ventilator assistance during Neurally Adjusted Ventilatory Assist (NAVA) to evaluate the effect of these on tidal volume, inspiratoy activity, comfort scales.

We propose to evaluate the ability to guide the titration according the patient's comfort scale. The intensity of the breathing sensations will be evaluated using the labeled visual analog scale (Banzett Scale).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Hospitalized in intensive care unit for an acute respiratory failure
* Intubated or tracheotomized and mechanically ventilated
* RASS score: 0;-2
* Weaning period

Exclusion Criteria:

* Hemodynamic instability
* Absence of consent
* Contraindication of nasogastric catheter insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of ventilatory comfort with the physiological parameters when varying the levels of pressure support and Neurally Adjusted Ventilatory Assist (NAVA) | 24hr
  To prove the feasibility of neurally adjusted ventilatory assist (NAVA) level titration according to the ventilatory comfort felt by the patient. The ventilatory comfort will be evaluated using the labeled visual analog scale (Banzett scale).

SECONDARY OUTCOMES:
Efficiency | 24hr
  The efficiency will be evaluated by using minute ventilation
Efficiency | 24hr
  The efficiency will be evaluated using arterial PCO2.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas TERZI, MD-PhD, Principal Investigator — University Hospital, Caen; Frédéric Lofaso, MD-PhD, Principal Investigator — University Hospital, Garches
Locations (1):
- CHU de Caen, Caen, France